CLINICAL TRIAL: NCT00975741
Title: An Open-label, Comparative, Randomized, Parallel, Multicenter Study to Determine the Efficacy and Safety of Two Dry Powder Inhalers (DPIs) Used for the Application of Mometasone in the Treatment of Asthma
Brief Title: Efficacy and Safety of Two Dry Power Inhalers (DPIs) Used for the Application of Mometasone in the Treatment of Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mantecorp Industria Quimica e Farmaceutica Ltd. (Industry)
Responsible Party: Celso Pereira Sustovich, Medical Director, Mantecorp Industria Quimica e Farmaceutica Ltda.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASM/P/01/1
Record Dates: First submitted 2009-08-12; First posted 2009-09-11 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Asthma
Keywords: Asthma; Mometasone furoate; Inhalation devices; Forced expiratory volume
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monodose device (Experimental): Mometasone furoate 400 µg DPI capsules administered through a monodose device.
  Interventions: Device: OXIMAX
- Multidose device (Active Comparator): Mometasone furoate 400 µg DPI capsules administered through a multidose device
  Interventions: Device: ASMANEX TWISTHALER

INTERVENTIONS:
Device: OXIMAX
  Arms: Monodose device
Device: ASMANEX TWISTHALER
  Arms: Multidose device

SUMMARY:
Mometasone furoate (MF) is a new potent synthetic corticosteroid. Internationally, MF is administered by a breath-actuated DPI and supplied in multidose devices. Capsules to be administered through a monodose device that would offer an alternative to MF DPI multidose treatment in terms of cost-effectiveness were developed in Brazil. The aim of the present non-inferiority clinical study was to evaluate both devices in terms of efficacy and safety.

DETAILED DESCRIPTION:
Background: Internationally, MF is administered by a breath-actuated DPI and supplied in multidose devices. Capsules to be administered through a monodose device that would offer an alternative to MF DPI multidose treatment in terms of cost-effectiveness were developed in Brazil. Results of laboratory analysis for respirable fraction, content uniformity of emitted dose and of the bulk powder and for percentage of particles < 1 micra of both MF 200 µg and MF 400 µg capsules have indicated their equivalent performance in comparison to MF DPI multidose.

Aim: The aim of the present non-inferiority clinical study was to evaluate both devices in terms of efficacy and safety.

Methods: Ninety-seven adult patients with moderate persistent asthma were randomized in two groups to receive for 60 days a dose of 400 µg of DPI MF once daily (at evening) using multidose or monodose device. Follow-up visits were scheduled at Days 7, 14, 28, 42 and 56. Efficacy was assessed by means of pulmonary function tests (spirometry - FEV1 and PEFR) at each visit. In addition, subjects have recorded twice daily PEFR, symptom scores and use of rescue medication throughout the study. Response to therapy was also assessed. Safety evaluations included monitoring of adverse events, vital signs, clinical laboratory tests (plasma cortisol concentrations were assessed at enrollment and repeated after 60 days of MF treatment; cortrosyn test was performed at the enrollment and after 60 days of MF treatment), and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of asthma for at least 6 months
* Baseline FEV1 must be > = 55% and < = 85% of predicted
* Increase in absolute FEV1 of >12%, with an absolute volume increase of at least 200 mL after reversibility testing
* Use of an adequate form of birth control by non-pregnant women of childbearing potential
* Absence of use of the following medication prior to the inclusion:

  * Beta 2 agonist short-acting (inhaled, oral)-12 Hours
  * Beta 2 agonist long-acting (inhaled)-48 Hours
  * Ipratropium bromide-12 hours
  * Cromolyn sodium, nedocromil-07 days
  * Astemizole-03 months
  * Cetotifeno-03 months
  * Another investigational drug-01 month
  * Theophyline-2 weeks
  * Antihistamines-07 days
  * Anticholinergics-07 days
  * Leukotriene modifiers-2 weeks
  * Oral decongestant long-acting-72 hours
  * Oral decongestant short-acting-24 hours

Exclusion Criteria:

* Women who were pregnant, breast-feeding, or are pre-menarcheal.
* Subjects who have used any investigational drug within the last 30 days
* Subjects who were receiving immunotherapy
* Subjects requiring the use of >12 puffs per day of Salbutamol on any 2 consecutive days
* Smokers or ex-smokers
* Subjects who are allergic to corticosteroids or beta-agonists
* Subjects who have required inpatient hospitalization for asthma control within the previous 3 months
* Subjects who have required ventilator support for respiratory failure secondary to their asthma within the last 5 years
* Subjects who have been treated in the emergency room (for a severe asthma exacerbation), or admitted to the hospital for management of airway obstruction, on two or more occasions within the last six months
* Subjects with clinical evidence of emphysema, chronic bronchitis, bronchiectasis, or cystic fibrosis
* Subjects with a significant history of renal, hepatic, cardiovascular, metabolic, neurologic, hematological, respiratory, gastrointestinal, cerebrovascular, or other significant medical illness or disorder which, in the judgment of the investigator, could have interfered with the study, or required treatment which might have interfered with the study
* Subjects who have experienced an upper or lower respiratory tract infection (viral or bacterial) within the previous 2 weeks prior to enrollment
* Subjects who have clinically significant abnormalities on chest x-ray at the Screening Visit or within the previous year
* Subjects who are known to be HIV positive
* Subjects who are known to be illicit drug abusers
* Subjects with hypothalamic-pituitary-adrenal (HPA) axis disturbances
* Subjects with severe pulmonary airflow obstruction showing to be life-threatening characterized by cyanosis, confusion, somnolence, coma or tiredness, thorax silent to hearing or showing weak respiration,PEFR <25% of the predicted normal, bradycardia (heartbeats bellow 60 beats per minute)
* Subjects with baseline FEV1 < 55% of the predicted normal
* Subjects with uncontrolled hypertension
* Subjects with suspected pneumonia, pneumothorax, pneumomediastinum, pulmonary tuberculosis, alpha-1 anti-trypsin deficiency, lung mycosis (blastomycosis, histoplasmic) or pulmonary cystic fibrosis
* Subjects with history of thoracic surgery or any previous malignancy of the lung
* Subjects with significant heart disease (e.g., previous acute myocardial infarction, angina pectoris, pulmonary edema or other cardiovascular disease which is characterized as life-threatening
* Subjects receiving beta-adrenergic blocking agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2002-10; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Difference in Forced Expired Volume in one second (FEV1) and Peak Expiratory Flow Rate (PEFR) measured by spirometry; number of puffs/day of rescue medication (Salbutamol) used by the subjects. | 56 days after initiation of therapy

SECONDARY OUTCOMES:
PEFR daily measurements, daily scores for asthma symptoms, response to therapy made by the Investigator, safety (hypothalamic-pituitary-adrenal axis evaluation and clinical laboratory measurements) and tolerability (adverse events). | 56 days after initiation of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Alberto C Pereira, MD, PhD, Principal Investigator — Hospital do Servidor Público Estadual, São Paulo
Locations (5):
- Brazil (5):
  - Hospital Universitário da Universidade Federal de Juíz de Fora, Juíz de Fora, Minas Gerais
  - UNIRIO, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Hospital do Servidor Público Estadual, São Paulo, São Paulo
  - Hospital Heliópolis, São Paulo, São Paulo

REFERENCES:
- [Derived] Pereira CA, Vianna FF, Cukier A, Stelmach R, Oliveira JC, Carvalho EV, Gomes EP, Mayo SV, Chibante AM, Domingues CP. Efficacy and safety of two dry-powder inhalers for the administration of mometasone furoate in asthma patients. J Bras Pneumol. 2010 Jul-Aug;36(4):410-6. doi: 10.1590/s1806-37132010000400004. English, Portuguese. PMID 20835586